CLINICAL TRIAL: NCT00406016
Title: A Multi-center, Open-label, Cohort Study to Assess Feasibility, Acute Safety, Tolerability and Pharmacokinetics of 4 Dose Regimens of Continuous Intrathecal ATI355 Infusion and Two Regimen of Repeated Intrathecal Bolus Injections in Acute Spinal Cord Injury Paraplegic and Tetraplegic Patients
Brief Title: Acute Safety, Tolerability, Feasibility and Pharmacokinetics of Intrath. Administered ATI355 in Patients With Acute SCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CATI355A2102
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2011-11

CONDITIONS: Acute Spinal Cord Injury
Keywords: Acute spinal cord injury;

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ATI355

INTERVENTIONS:
Drug: ATI355

SUMMARY:
This study will evaluate the acute safety, tolerability, feasibility and pharmacokinetics of 6 dose regimens of ATI355 in acute spinal cord injury patients

ELIGIBILITY:
Inclusion criteria

* Acute spinal cord injury paraplegic and tetraplegic patients with confirmed classification of ASIA A (C5 ≤ lesion ≤ T12; 4-14 days post-injury (i.e. study drug treatment must begin 4-14 days post injury) for paraplegic patients and for those tetraplegic patients who do not require artificial respiration at time of treatment initiation within the 4-14 days time interval. In those tetraplegic patients who still require artificial respiration in the 4-14 days time interval treatment can be initiated up to 60 days post-injury as soon as the patient is weaned off the respiratory machine.)
* Tetraplegic patients who were initially diagnosed as ASIA A (neurologically complete lesion) at screening and turned into ASIA B (neurologically incomplete lesion) at baseline.
* Hemodynamically stable (at baseline).
* For female patients of child bearing potential, written agreement to abstain from intercourse during the first 12 weeks of the study and then subsequent use of a double-barrier local contraception, i.e. intra-uterine device plus condom, or spermicidal gel plus condom for up to one year post study drug treatment. Patients must receive documented counseling on contraceptive measures.
* For Cohort 5: Acute spinal cord injury tetraplegic patients with confirmed classification of ASIA A: Cervical lesions (C5 ≤ lesion ≤ T1). 4-28 days post-injury (i.e. study drug treatment must begin 4-28 days post injury). Tetraplegic patients who are allowed to start treatment are those who either do not require mechanical ventilation or who do not completely depend on mechanical ventilation but show some degree of spontaneous ventilation. Only those modes of ventilation where the patient must initiate all breaths are allowed (e.g. continuous positive airway pressure [CPAP]).

Exclusion criteria

* Complete anatomical transection confirmed by MRI or trauma caused by ballistic or other injury that directly penetrates the spinal cord including gunshot and knife wounds.
* Magnetic Resonance Imaging (MRI) indicating complete obstruction of the intrathecal space.
* Presence of one of the following:
* multiple spinal cord lesions
* cauda equina damage
* major brachial or lumbar plexus damage/trauma
* significant head trauma (e.g. cortical damage/lesion), or other injury that was, in the opinion of the investigator, sufficient to interfere with the assessment of the spinal cord function or otherwise compromise the validity of the patient's data.
* Other significant preexisting or current systemic disease such as lung, liver (exception: history of uncomplicated Hepatitis A), gastrointestinal, cardiac, immunodeficiency (including human immunodeficiency virus [HIV]) or kidney disease; or active malignancy or any other condition as determined by history or laboratory investigation that could cause a neurological deficit including syphilis, myelopathy, clinically relevant polyneuropathy, etc.
* History of meningitis, meningoencephalitis, epilepsy or life-threatening allergic or immune-mediated reaction.
* History of or current autoimmune disease or an acute episode of Guillain-Barre syndrome.
* Patients with uncontrolled bleeding diathesis and/or on concomitant treatment with coumarin anticoagulant.
* Presence of any unstable medical or psychiatric condition (defined by the Diagnostic and Statistical Manual of Mental Disorders-IV [DSM-IV]) that could reasonably have been expected to subject the patient to unwarranted risk from participation in the study or result in a significant deterioration of the patient's clinical course.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/ml).
* Hemoglobin levels below 8.0 g/dl and/or patients who required greater than 10 (ten) blood transfusions since the acute injury
* Patients with concomitant treatment with Metamizole from Screening until end of Follow Up phase
* Mechanical ventilation will be allowed for patients in Cohort 5, the patient must not depend completely on the ventilation but should show some degree of spontaneous ventilation. Only those modes of ventilation where the patient must initiate all breaths are allowed (e.g. continuous positive airway pressure [CPAP]).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Feasibility, Safety and Tolerability of a continuous intrathecal (i.t.) infusion or i.t. repeated bolus injections of ATI355 in patients with acute spinal cord injury at every visit and Assessment of serum and CSF pharmacokinetics at predefined visits. | 1 year

SECONDARY OUTCOMES:
Immunogenicity of ATI355 in acute spinal cord injury patients up to one year. | 1 year
Early potential signal of efficacy by the American Spinal Cord Injury Association (ASIA) protocol and pharmacodynamic changes assessed by electrophysiology tests for up to one year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Canada (4):
  - Novartis Investigative site, Calgary
  - Novartis Investigative site, Montreal
  - Novartis Investigative site, Toronto
  - Novartis Investigative site, Vancouver
- Germany (9):
  - Novartis Investigative site, Bad Wildungen
  - Novartis Investigative site, Bayreuth
  - Novartis Investigative site, Bochum
  - Novartis Investigative site, Hamburg
  - Novartis Investigative site, Heidelberg
  - Novartis Investigative site, Karlsbad-Lagensteinbach
  - Novartis Investigative site, Murnau am Staffelsee
  - Novartis Investigative site, Tübingen
  - Novartis Investigative site, Ulm
- Novartis Investigative site, Zurich, Switzerland